CLINICAL TRIAL: NCT03363074
Title: Comparison of the Effects of Low-Level Therapy Laser and Orthotic Insole on Pain, Function and Muscle Strength in Subjects With Stage 1-2 Tibialis Posterior Tendon Insufficiency: Randomized Study
Brief Title: Low-Level Laser Therapy and Orthotic Insole in Tibialis Posterior Tendon Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Cansu Koltak, Research Assistant, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETK00-2017-0204
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Posterior Tibial Tendon Insufficiency
Keywords: Low-Level Laser Therapy, Orthotic Insoles
MeSH Terms: conditions — Posterior Tibial Tendon Dysfunction | interventions — Foot Orthoses; Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orthotic Insole (Experimental): Device: Orthotic Insole 8-week follow-up with Orthotic Insole
  Interventions: Device: Orthotic Insole
- Low-level Laser Therapy (Experimental): Low-Level Laser 5-week follow-up
  Interventions: Device: Low-Level Laser

INTERVENTIONS:
Device: Orthotic Insole — A computer numerical control machine was used to product insoles according to pedobarographic pressure data;35 Shore A hardness ethyl vinyl acetate was used for the main insole,and 3mm,15 Shore A hardness ethyl vinyl acetate was used for covering.Orthotic insoles have been emplemented in a pair of sports shoes.
  Arms: Orthotic Insole
Device: Low-Level Laser — A low density laser with a power density of 0.05-0.10 (w / cm2), a therapeutic dose of 0.7-7 (j / cm 2) of gallium-arsenic 904 nm will be applied. It will be 3 administered times a week for 5 weeks. Laser treatment will be applied along the tibialis posterior tendon. 3 different point (proximal tibial tendon, distally tibial tendon and posterior medial malleol) applications will be done.
  Arms: Low-level Laser Therapy

SUMMARY:
The purpose of this study is to compare low-level laser therapy and insole interventions on pain, function and muscle strength in subjects with posterior tendon insufficiency.

DETAILED DESCRIPTION:
Purpose of the research; stage 1-2 tibialis between the ages of 18-60 is a comparison of low-level laser therapy and orthotic insole on pain, function and muscle strength in subjects with posterior tendon insufficiency.

Type of research:

This study is a randomized comparative intervention study.

Place to do research:

The study will be carried out in the Prosthetic Orthotics and Biomechanics Center of the Department of Physiotherapy and Rehabilitation of the Faculty of Health Sciences of the Eastern Mediterranean University.

Evoluotion and Sample Size Of Research:

Subjects aged 18-60 who volunteered by the physician from Eastern Mediterranean University who had been diagnosed with tibialis posterior insufficiency would be included in the study.According to the power analysis using G-Power program; a total of 52 subjects will be included in the calculation of Cohen d = 0.8, α = 0.05, β = 0.20, assuming that the nonparametric Mann Whitney-U test is used for comparison between the two groups. It was decided that 60 people would be taken from the survey without a 20% loss.

Volunteers Including / Exploring Criteria:

Inclusion Criteria:

* Taking the diagnosis of stage 1 - 2 tibialis posterior insufficiency by the physician,
* Be between the ages of 18 and 60,
* The absence of a different orthopedic or neurological disease that may affect the lower extremity biomechanics,
* Not having a systemic disease that keeps feet. Having not received any treatment from the foot area in the last 1 year.

Exclusion Criteria:

* Having lower extremity discrepancy more than 1 centimeter (cm),
* Having no ambulation without help.

Reserch Method:

Our study consists of two groups and the subjects will be taken to these groups using a random number table. One group of our study is a and orthotic insole group and the other group is a low -level laser therapy group. The orthotic insole group will use their special insoles for 8 weeks. The low-level laser therapy group will receive treatment at the Prosthesis Orthotic Biomechanics Center of the Eastern Mediterranean University three times a week for 5 weeks. Laser will be applied along the tibial posterior tendon. Before the data is collected, the individual will be informed about the equipment to be used in the tests. There will be 1 trial before assessment and treatment so that participants can become familiar with the equipment. All assessments and insoles will be applied by the same physiotherapist.

Data Collection Vehicles and Properties:

To be applied to the patient:

1.Pain Assessment ; with digital algometer 2.Muscle strength assessment ; with Isokinetic Dynamometer 3.Evulation of Foot Function ; with Foot Function Index 4.Other Assessment ; Foot Posture Index, International Physical Activity Index(short form)

1. Pain Assessment ; It will be assessed with pain algometer. Before starting treatment, measurements will be taken at three different points of the tibialis posterior tendon. Three measurements from each point will be taken. The right and left foot will be evaluated. the previously assessed regions will be reevaluated at the end of the treatment.
2. Muscle strength assessment Using the isokinetic dynamometer (Humac Norm Isocynetic Dynanometer), the force values of the inverter and the evertor muscles of the foot will be measured.Before starting the test, a standard warm-up program will be applied for 3 minutes without resistance in the patient bicycle ergometer. At the same time, passive stretching of the patients' gastrocnemius and soleus muscles. Subjects movements will be evaluated at 10 repetitions at 180º / sec, 10 repetitions at a rate of 240º / sec. Before each angular velocity, subjects are allowed to perform 3 repeated trials and after 10 seconds rest, tests will be applied. Unilateral measurement will be performed.
3. Evulation of Foot Function ; with Foot Function Index. This scale evaluates the severity of foot pain in different situations. It consists of 3 subtitles and contains 23 questions in total. Turkish version adaptation study is done, valid and reliable measure. Each question takes between 0 and 10 points. the total score is divided by the number of questions answered and scaled by finding the value over 100.
4. Other Assessment;

   1. Foot Postüre Index : Index will be used to determine the flat foot of the individuals. According to the scale, a total score of -12 to +12 is obtain with a score under six headings during static standing. Medial longitudinal arch height increases with increasing points, medial longitudinal height decreases with increasing points. Our study will include individuals who have received a minimum score of +6 as in similar research.
   2. International Physical Activity Index (short form) (IPAQ) : The index will be used to determine the physical activity levels of individuals. With the scale of Turkish validity and reliability studies, low, medium and high intensity activity periods of the individuals in the last week will be evaluated under 7 questions and the average energy expenditure value will be obtained in kcal / week.Individuals will be asked to do this questionnaire on a regular basis every week.

Treatment Program:

Low-level Laser Therapy Group; A low density laser with a power density of 0.05-0.10 (w / cm2), a therapeutic dose of 0.7-7 (j / cm 2) of gallium-arsenic 904 nm will be applied. It will be administered 3 times a week for 5 weeks. Laser treatment will be applied along the tibialis posterior tendon. 3 different point applications will be done. Proximal tibial tendon, distally tibial tendon and medial malleoli posterior.

Orthotic Insole Group:

Individuals will be operated by pressing on a fixed pedobarograph (Medilogic, platform basic, Germany) embedded in a 5-m wooden floor and foot pressure measurements will be taken. Of the three successful measurements made, the one closest to the normal walk will be recorded. According to the foot pressure measurement, the MLA, TA and MTK attachments will be used in the insoles design developed by the modeling program.

The individual will use the insoles for 8 weeks with the appropriate footwear. individuals will be required to fill in the international physical activity scale each week. As well as how many hours a day each of his or her inviduals have been using their insoles. A table will be created and given to the individuals to write how many hours they are using.

ELIGIBILITY:
Inclusion Criteria:

* Taking the diagnosis of stage 1 - 2 tibialis posterior insufficiency by the physician,
* Be between the ages of 18 and 60,
* The absence of a different orthopedic or neurological disease that may affect the lower extremity biomechanics,
* Not having a systemic disease that keeps feet.
* Having not received any treatment from the foot area in the last 1 year.

Exclusion Criteria:

* Having lower extremity discrepancy more than 1 centimeter (cm),
* Having no ambulation without help.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-08-25 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
Change in Foot Function Assesed With Foot Function Index | Baseline and 6 week for Low-Level Laser Therapy Group - 8 week for Orthotic Insole Group
  This scale evaluates the severity of foot pain in different situations. It consists of 3 subtitles and contains 23 questions in total. Turkish version adaptation study is done, valid and reliable measure. The total score obtained by the patient between 0-10 of each question was scaled by obtaining a score of 100 with the number of answered questions

SECONDARY OUTCOMES:
Change in Muscle Strength Assesed With Humac Norm Isocynetic Dynanometer | Basline and 6 week for Low-Level Laser Therapy Group - 8 week for Orthotic Insole Group
  The force values of the inverter and the evertor muscles of the foot will be measured. Before starting the test, a standard warm-up program will be applied for 3 minutes without resistance in the patient bicycle ergometer. At the same time, passive stretching of the patient's gastrocnemius and soleus muscles. Subjects movements will be evaluated at 10 repetitions at 180º / sec, 10 repetitions at a rate of 240º / sec. Before each angular velocity, subjects are allowed to perform 3 repeated trials and after 10 seconds rest, tests will be applied. Unilateral measurement will be performed.
Change in Foot Pain Assesed With Digital Algometer | Baseline and 6 week for Low-Level Laser Therapy Group - 8 week for Orthotic Insole Group
  The pain from the three different points of the tendon with the sensor will be assessed. 3 different point (proximal tibial tendon, distally tibial tendon and posterior medial malleol.

CONTACTS AND LOCATIONS:
Overall Officials: Yasin Yurt, PhD, Principal Investigator — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Mersin, Famagusta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No